CLINICAL TRIAL: NCT01638481
Title: Determining the Chronology of Occult and Gross Coagulopathy in Thermally Injured Patients: A Systems Biology Approach
Brief Title: Chronology of Occult and Gross Coagulopathy in Burn Patients
Status: Completed | Type: Observational
Sponsor: Medstar Health Research Institute (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 58802-LS
Record Dates: First submitted 2012-07-09; First posted 2012-07-11 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Thermal Burns

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Group #1 - Burns affecting less than 10% BSA
- Group #2 - Burns affecting 10%-30% TBSA
- Group #3 - Burns affecting 31%-50% TBSA
- Group #4 - Burns affecting 51%-70% TBSA
- Group #5 - Burns affecting >70% TBSA

SUMMARY:
The purpose of the study is to identify the inflammatory and coagulation pathways and mechanisms that are activated immediately following burn injury, and how they affect outcomes in terms of organ failure and death. This study also addresses the limitation of current tests (PT, PTT, and platelet counts) employed to identify coagulation disturbances in severely injured patients both in a comprehensive and rapid manner.

ELIGIBILITY:
Inclusion Criteria:

* Patients, male or female, > or = 18 years of age, who arrive at Burn/Trauma Center with anticipated admission to The Burn Center within 4 hours of injury, with a thermal burn injury due to flash, flame, contact with hot object or liquid.

Exclusion Criteria:

* Patients suffering concomitant trauma that are in hemorrhagic shock. Patients with a preexisting history of coagulopathy, or currently taking anti-coagulants. Children and pregnant women. Patients with chemical or electrical injury. Patients who do not fluently speak either English or Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Burn injury patients will be enrolled in the study upon arrival at Trauma Center.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2021-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Shupp, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States